CLINICAL TRIAL: NCT00531336
Title: Comparison of Combined Therapy of Intravitreal Injection of Avastin and Macugen Versus Mono-Therapy The MAAM Study - a Pilot Study
Brief Title: MAAM Study: Avastin and Macugen Versus Avastin Versus Macugen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Susanne Binder Prof, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK06-001839-18
Record Dates: First submitted 2007-09-15; First posted 2007-09-18 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2008-10

CONDITIONS: Macular Degeneration
Keywords: age-related Macular degeneration; Macugen; Avastin
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab; pegaptanib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Avastin first followed by retreatment of Macugen
  Interventions: Drug: intravitreal injection of Bevacizumab (Avastin); Drug: Pegaptanib (Macugen)
- 2 (Active Comparator): Avastin intravitreally every 6 weeks
  Interventions: Drug: intravitreal injection of Bevacizumab (Avastin)
- 3 (Active Comparator): Macugen intravitreally every 6 weeks
  Interventions: Drug: Pegaptanib (Macugen)

INTERVENTIONS:
Drug: intravitreal injection of Bevacizumab (Avastin) — 1.25 mg Avastin intravitreally applied once in arm 1 every 6 weeks in arm 2
  Arms: 1; 2
Drug: Pegaptanib (Macugen) — 0.3 mg intravitreally applied every 6 weeks as long as required
  Arms: 1; 3

SUMMARY:
The first results of Anti-Vascular Endothelial Growth Factor (VEGF) therapy were very promising and superior to established therapies. Three different substances (all of them applied intravitreally) are available, but comparative studies have not yet been conducted. In this pilot study, the safety (number of adverse events) and efficacy (distance acuity testing retinal thickness measurement) of Avastin and Macugen applied as monotherapy will be compared to a combined treatment of Avastin followed by Macugen used for retreatment.

At least equal results of the combined therapy are expected.

DETAILED DESCRIPTION:
The role of Vascular Endothelial Growth Factor (VEGF) in the pathogenesis of neovascular diseases like choroidal neovascularization (CNV) and proliferative diabetic retinopathy has been demonstrated in a series of publications. Therefore intravitreally applied VEGF antagonists have been used in the treatment of CNV in age-related macular degeneration (AMD) and diabetic cases. Three anti-VEGFs are available: Macugen® (Pegaptanib), Avastin® (Bevacizumab) and Lucentis® (Ranibizmab). Pegaptanib sodium is an aptamer designed to bind the VEGF 165 isoform with high affinity. Bevacizumab is a humanized monoclonal antibody to VEGF designed for intravenous administration and approved for the treatment of colorectal cancer. Ranibizumab is an anti-body binding site fragment that is derived from the same anti-VEGF antibody as bevacizumab. The decrease of retinal thickness measured in the OCT provides information concerning the amount of intraretinal fluid accumulation and therefore for the activity of a neovascular lesion. It has been proven that the aqueous humor levels of VEGF of eyes with CNV are significantly higher than those of eyes without ocular or systemic diseases. The retinal thickness and the VEGF concentration in the aqueous humor should give a good correlation to the anti vasogenic effect of the intravitreal treatment. In this study bevacizumab and pegaptanib as monotherapy should be compared with a combined therapy of bevacizumab applied first with pegaptanib used for retreatment. The benefit of this combined therapy should be that an initial blockage of all VEGF isoforms is necessary whereas for retreatment the blockage of the most important isoform in the pathogenesis of CNV is sufficient and the normal function of the retinal pigment epithelium and the choriocapillaris is not affected.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Predominantly occult CNV
* Greatest diameter of the lesion < 5400µm
* Distance acuity > 0.1

Exclusion Criteria:

* Complicating general disorders inflicting with healing process
* Vision threatening diseases other than CNV
* Prior treatment for CNV
* Ophthalmic surgery within 4 weeks
* Not consented patients

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
retinal thickness | 54 weeks

SECONDARY OUTCOMES:
distance acuity | 54 weeks
number of adverse events | 54 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Krebs, MD, Principal Investigator — Ludwig Boltzmann Institute for Biomicroscopic Lasersurgery
Locations (1):
- Ludwig Boltzmann Institute for Retinology and Biomicroscopic Lasersurgery, Vienna, Vienna, Austria